CLINICAL TRIAL: NCT04401995
Title: Randomized Neoadjuvant Pilot Phase II Study of TLR9 Agonist Vidutolimod (CMP-001) in Combination with Nivolumab Vs. Nivolumab in Stage IIIB/C/D Melanoma Patients with an Integrated Imaging Biomarker
Brief Title: Study of TLR9 Agonist Vidutolimod (CMP-001) in Combination with Nivolumab Vs. Nivolumab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Diwakar Davar (Other)
Collaborators: Checkmate Pharmaceuticals (Industry); CellSight Technologies, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Diwakar Davar, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HCC 20-049
Record Dates: First submitted 2020-05-18; First posted 2020-05-26 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Melanoma
Keywords: residual volume of tumor (RVT); standard uptake value (SUV)
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nivolumab and Vidutolimod (CMP-001) Combination with [18F]F-AraG PET/CT (Experimental): Prime Phase - Nivolumab 240mg IV, every 2 weeks starting with Cycle 2 (Cycles 2,4,6) for 6 weeks in combination with Vidutolimod 5mg subcutaneous 1st dose, and the remaining injections, 10mg intra-tumorally will be administered Weeks 2-7. [18F]F-AraG PET/CT, single bolus injection of 5 (±10%) mCi IV into a vein, Screening and at Week 2.
  Boost Phase - Nivolumab 480mg IV, every 4 weeks and CMP-001 5mg subcutaneous every 4 weeks up to 48 weeks.
  Interventions: Drug: Vidutolimod (CMP-001); Biological: Nivolumab; Other: [18F]F-AraG PET/CT
- Nivolumab with [18F]F-AraG PET/CT (Experimental): Prime Phase - Nivolumab 240mg IV, every 2 weeks starting with Cycle 2 (Cycles 2, 4, 6) for 6 weeks. [18F]F-AraG PET/CT, single bolus injection of 5 (±10%) mCi IV into a vein, Screening and at Week 3.
  Boost Phase - Nivolumab 480mg IV, every 4 weeks starting from the time of surgery recovery for up to 48 weeks.
  Interventions: Biological: Nivolumab; Other: [18F]F-AraG PET/CT

INTERVENTIONS:
Drug: Vidutolimod (CMP-001) — A molecule comprised of a 30 nucleotide strand, flanked by 10 guanines on either end. The nucleotide strand is surrounded by a Qβ viral-like protein. The intended mechanism of action of CMP-001 in oncology is the activation of TLR9 in pDC within the tumor or the tumor-draining lymph nodes (tumor-associated pDC).
  Arms: Nivolumab and Vidutolimod (CMP-001) Combination with [18F]F-AraG PET/CT
Biological: Nivolumab — a fully human Ig G4 antibody that blocks PD-1. Nivolumab was initially approved by the FDA for the treatment of patients with unresectable or metastatic melanoma and disease progression following ipilimumab and, if BRAF V600 mutation positive, a BRAF inhibitor. Nivolumab has also been FDA approved to treat patients with advanced squamous non-small cell lung cancer (NSCLC) with progression on or after platinum-based chemotherapy, as well as advanced renal cell carcinoma.
Other: [18F]F-AraG PET/CT — [18F]F-AraG is an 18F-labeled analog of arabinofuranosylguanine (AraG), a compound that has shown remarkably selective accumulation in T cells. It has several advantages over conventional [18F] and existing small molecule PET agents being investigated for immuno-monitoring. [18F]F-AraG has lower accumulation and more efficient efflux from cancer cells than a dCK agent.

SUMMARY:
The main goal of this research study is to determine how nivolumab and nivolumab/Vidutolimod (CMP-001) combination affect the likelihood of destroying melanoma involving lymph node and/or in-transit/satellite areas.

The main goal of the PET/CT scan with 18F]F-AraG is to evaluate how [18F]F-AraG uptake changes before and after administration of either nivolumab or nivolumab/CMP-001 combination.

DETAILED DESCRIPTION:
This is a phase II pilot study designed to compare the pCR rate of two neoadjuvant immunotherapies in high-risk resectable melanoma with two integrated biomarkers. The integrated [18F]F-AraG imaging biomarker images activated CD8+ T cells. The CD8+ T cell density biomarker quantitates CD8+ T Cells using an automated method. The primary purpose of the study is to describe the correlation between pCR and the distribution of either biomarkers in patients receiving either neoadjuvant Vidutolimod (CMP-001)/nivolumab or neoadjuvant nivolumab.

Patients with stage IIIB-IIID cutaneous (or unknown primary) melanoma with palpable nodal disease who have yet to undergo definitive surgery are eligible to enroll. Patients with nodal relapse including those who have received prior adjuvant IFN and/or ipilimumab are eligible to enroll.

Suitable patients will be identified pre-operatively. Patients will undergo a 28 day screening evaluation including surgical assessment, clinical assessment, systemic/CNS staging scans, and laboratory studies to confirm suitability. Patients will undergo biopsies of both planned injected and uninjected lesions (Arm A) and target lesion (Arm B). Biopsies of these lesions will occur pre-treatment, at W3 or W4 and the target lesion(s) will be resected at the time of surgery.

Eligible patients will be randomized 1:1 to receive Arm A (neoadjuvant Nivolumab/(CMP) vs. Arm B (neoadjuvant Nivolumab) during the (Prime Phase) pre-operatively. Patients randomized to Arm A will receive: Nivolumab 240mg IV q2 x3 and CMP-001 5mg SC 1st dose then 10mg IT 2nd-7th doses (7 weeks). Patients randomized to Arm B will receive: Nivolumab 240mg IV q2 x3 (6 weeks).

[18F]F-AraG PET-CT scan (18-F PET) is an integrated biomarker and will be performed at 2 imaging time-points: pre-treatment (pre-W1) and on-treatment (W2). At each imaging timepoint, [18F]F-AraG will be administered by a licensed nuclear medicine technologist under the supervision of a nuclear medicine physician on an outpatient basis. Each patient will receive a single bolus injection of 5 mCi [18F]F-AraG IV into a hand or arm vein. At Screening and W2 imaging timepoints, following [18F]F-AraG injection, a 30-min static PET-CT scan will be performed covering the brain to the upper legs.

For CD8+ T cell density assessments, patients will undergo biopsies at 2 timepoints: pre-treatment (Screening) and on-treatment (W3 or W4). In Arm A, patients will undergo biopsies of planned injected and a 2nd uninjected lesion. At each imaging timepoint, biopsies will be performed.

Following the Prime Phase and restaging systemic scans, patients will undergo surgical resection.

Post-operatively, patients will continue to receive maintenance therapy (Boost Phase) per randomization. In the Boost Phase, patients randomized to Arm A (neoadjuvant Nivolumab/(CMP) will receive 480mg IV q4 x12 along with Vidutolimod (CMP-001) 5mg SC q4 x12 over a 48 week period; while patients randomized to Arm B (neoadjuvant Nivolumab) will receive Nivolumab (480mg IV q4 x12 over a 48 week period). In the post-operative period, CMP-001 will be administered subcutaneously (Arm A only).

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the study.
2. Be ≥ 18 years of age on day of signing informed consent.
3. Willingness to undergo [18F]F-AraG PET imaging at pre- and week 3 timepoints.
4. Diagnosis of histologically or cytologically confirmed diagnosis of cutaneous melanoma belonging to one of the following AJCC TNM stages:

   1. Tx or T1-4 and
   2. N1b, or N1c, or N2b, or N2c, or N3b, or N3c and
   3. M0

   Patients are eligible for this trial either at presentation for primary melanoma with concurrent regional nodal metastasis; or at the time of clinical detected nodal recurrence; and may belong to any of the following groups:
   * Primary cutaneous melanoma with clinically apparent regional lymph node metastases.
   * Clinically detected recurrent melanoma at the proximal regional lymph node(s) basin.
   * Clinically detected primary cutaneous melanoma involving multiple regional nodal groups.
   * Clinical detected nodal melanoma (if single site) arising from an unknown primary.
   * In-transit and/or satellite metastases with regional lymph node involved permitted if considered potentially surgically resectable at baseline.
   * NOTE: Patients whose sole site of disease is regional lymph node involvement of the parotid LN basin are not eligible for this neoadjuvant study.
   * NOTE: Patients with only in-transit and/or satellite metastases without regional lymph node involvement are not eligible for this neoadjuvant study.
   * NOTE: Determination of potential resectability must be made at baseline to be eligible for this neoadjuvant study.
   * NOTE: Patients with mucosal and/or uveal melanoma are not permitted to enroll. Patients with melanomas of unknown primary may be enrolled at the discretion of the treating investigator in discussion with Principal Investigator.
5. Presence of injectable and measurable disease based on RECIST 1.1.
6. Willing to undergo tumor biopsy (core, punch, incisional or excisional). Patients must undergo biopsy (core, punch) or open biopsy (incisional, excisional) within 4 weeks of registration on the study and at W4-5.
7. Performance status of 0 or 1 on the ECOG Performance Scale.
8. Demonstrate adequate organ function as defined below performed on screening labs obtained within 4 weeks of registration.

   * Absolute neutrophil count (ANC) ≥1,500 /mcL
   * Hemoglobin ≥9 g/dL or ≥5.6 mmol/L
   * Platelets ≥100,000 / mcL
   * Serum creatinine or Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN.
   * Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN.
   * AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN.
   * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
   * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
9. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 26 weeks after the last dose of study medication (Section 5.7.2). Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
11. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 26 weeks after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. History of uveal or mucosal melanoma.
2. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
4. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
   * Note: Subjects with autoimmune disorders of Grade 4 while on prior immunotherapy will be excluded. Subjects who developed autoimmune disorders of Grade ≤ 3 may enroll if the disorder has resolved to Grade ≤1 and the subject has been off systemic steroids at doses >10 mg/d for at least 2 weeks.
5. Active (i.e., symptomatic or growing) central nervous system (CNS) metastases.
6. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
7. Has a systemic disease that requires systemic pharmacologic doses of corticosteroids greater than 10mg daily prednisone (or equivalent). Subjects who are currently receiving steroids at a dose of ≤10mg daily do not need to discontinue steroids prior to enrollment Subjects that require topical, ophthalmologic and inhalational steroids would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study. Subjects who require active immunosuppression (greater than steroid dose discussed above) for any reason are excluded.
8. Has evidence of interstitial lung disease or active, non-infectious pneumonitis.
9. Has an active infection requiring systemic therapy.
10. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
11. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
12. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 26 weeks after the last dose of trial treatment.
13. Has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137 or BRAF/MEK inhibitor. Prior treatment with ipilimumab or interferon alfa is allowed. Patients with history of allergic or hypersensitivity reaction to interferon alfa or ipilimumab are also excluded.
14. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
15. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected. Patients with treated Hepatitis B/C with no evidence of active infection may be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Major Pathologic Response Rate (MPR) | At the time of surgery (Week 8-10)
  A ratio of responders (to treatment) to total number of tumors (responders plus non-responders to treatment). Immune-related pathologic response rate based on the percent (%) of residual volume of tumor (RVT). Pathologic Non Response (pNR) is defined as %RVT>50%; Partial Pathologic Response (pPR) is defined as 10%< %RVT<50% (at least 10%, up to 49%); Major Pathologic Response (MPR) is defined as %RVT≤10%; Pathologic
Pathologic Complete Response (pCR) Rate | At the time of surgery (Week 8-10)
  Per Immune-related pathologic response criteria (irPRC), pCR is defined as 0% RVT remaining in post-therapy specimen.
Distant-metastasis free survival (DMFS) | At 6-months, 12-months, 2-year, 3-year, 5-year; up to 5 years
  The length of time from initiation of treatment until distant-metastasis of melanoma or death.

SECONDARY OUTCOMES:
Tumor PET response via [18F]F-AraG | At Week 1 (baseline) and Week 5
  [18F]F-AraG is an experimental PET imaging agent. Tumor PET response will be assessed via standard uptake values (SUV) measured as SUVmax, SUVpeak, SUVmean, and SUVtotal.The max, peak, mean and total values for each patient will be used to determine the average standard uptake values for the study population. The possible range of SUV values is between 0 - 100. Higher SUV correlates with greater malignancy.
Relapse-Free Survival (RFS) | At 6-months, 12-months, 2-year, 3-year, 5-year; up to 5 years
  The length of time from initiation of treatment until melanoma relapse or death.
Overall Survival (OS) | At 6-month, 12-months, 2-year, 3-year, 5-year; up to 5 years
  The length of (survival) time from the start of treatment until death from any cause.
Adverse Events at Least Possibly Related to Study Treatment | Up to 5 years
  Toxicities defined by NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 are adverse events classified as either possibly, probably, or definitely related to study treatment. The maximum grade for each type of toxicity will be recorded and the frequency of toxicities will be tabulated for the study population.

OTHER OUTCOMES:
CD8+ T cell density | Pre-treatment (Screening), at Week 3 of treatment; up to 21 days
  The quantity of CD8 + T-cells that infiltrate tumors, measured via flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: Diwakar Davar, MD, M.Sc, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No